CLINICAL TRIAL: NCT02434575
Title: ROPE Registry Project to Determine the Safety and Efficacy of Prostate Artery Embolisation (PAE) for Lower Urinary Tract Symptoms Secondary to Benign Prostatic Enlargement (LUTS BPE)
Brief Title: UK ROPE Register Study
Acronym: UK ROPE
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: British Society of Interventional Radiologists (Unknown); British Association of Urological Surgeons (Unknown); National Instutite of Health and Care Excellence (Unknown)
Responsible Party: Principal Investigator, Dr Grace Carolan-Rees, Cedar Director, Cardiff and Vale University Health Board
Other Study IDs: 14/NE/0128
Record Dates: First submitted 2015-03-20; First posted 2015-05-05 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Lower Urinary Tract Symptoms; Prostatic artery embolisation; Transurethral resection of the prostate; Benign prostatic hyperplasia; Benign prostatic enlargement
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PAE: Men with LUTS BPE who have opted for PAE at a participating site, and have consented to take part in the UK ROPE Register Study.
- TURP: Men with LUTS BPE who have consented to TURP at a participating site, and have consented to the UK ROPE Register Study.
- Other: Men with LUTS BPE who have had an Open Prostatectomy or laser surgery at a participating site, and have consented to the UK ROPE Study.

SUMMARY:
This registry study enables us to collect data on the treatment of LUTS using prostate artery embolisation (PAE), and other surgical methods to answer the following questions posed by NICE in 2013:

* Is PAE a safe and effective treatment option for LUTS caused by prostate enlargement?
* How does PAE compare with conventional surgical treatments? This will primarily be a surgical procedure called transurethral resection of the prostate (TURP) (see below).
* Which patients would most benefit from PAE over the other treatment options?

DETAILED DESCRIPTION:
This is a study protocol for the UK ROPE Register for Lower Urinary Tract Symptoms (LUTS). This register enables us to collect data on the treatment of LUTS using prostate artery embolisation (PAE), and other surgical methods to answer the following questions posed by NICE in 2013:

* Is PAE a safe and effective treatment option for LUTS caused by prostate enlargement?
* How does PAE compare with conventional surgical treatments? This will primarily be a surgical procedure called transurethral resection of the prostate (TURP) (see below).
* Which patients would most benefit from PAE over the other treatment options? This study involves populating the UK ROPE Register with data from patients who have undergone prostate artery embolisation (PAE) and the current standard treatment in the UK, transurethral resection of the prostate (TURP). All consecutive patients receiving PAE in UK sites taking part in this study over the course of 12 months (from the date that the first patient is enrolled) will be invited to join the UK ROPE register. At least 150 PAE patients will be enrolled into this study, and a comparable number of TURP patients (at least 150 patients also) from a maximum of 18 sites in the UK. It is anticipated that each site will enrol between 10 and 30 PAE patients in 12 months. Enrolment will only continue past 12 months until 150 PAE patients have been added to the register.

NICE has suggested keeping a registry or database of patients who have undergone this procedure in the UK. so that we can find out more about how safe and effective it is for patients and how it compares to the other established treatments available such as surgery. The UK ROPE Register will be owned and hosted by the British Society of Interventional Radiologists (BSIR) and the British Association of Urological Surgeons (BAUS). The register will be built by Dendrite, a commercial company that specialise in making medical registers and databases. Cedar, a consortium of Cardiff & Vale UHB and Cardiff University and an External Assessment Centre (EAC) to NICE, was commissioned to facilitate the registry research. Cedar's role is to work with the steering group (consisting of BSIR, BAUS, and NICE representatives) to help build the ROPE Register and ensure that the right data points are collected to answer research questions for NICE. Cedar will also perform the data analysis from the ROPE Register and will publish the results in a peer-reviewed scientific journal.

ELIGIBILITY:
Inclusion Criteria:

* Men with LUTS who have consented for PAE, TURP, open prostatectomy or laser surgery at a participating site
* Able to read, write and understand English
* Capable of giving informed written consent

Exclusion Criteria:

* Not able to read, write or understand English
* Not able/willing to provide informed written consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men with LUTS BPE who have consented to PAE, TURP, Open prostatectomy or laser surgery at a participating UK site.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
IPSS change for PAE patients, from baseline 12 months post procedure | 12 months
  Comparison of IPSS questionnaire score at baseline at 12 months post-PAE procedure

SECONDARY OUTCOMES:
IPSS comparison of PAE with TURP, 12 months post-procedure | 12 Months
  Comparison of IPSS score changes between PAE and TURP cases, 12 months post-procedure. Non inferiority study.
Safety of PAE procedure - Number of patients with adverse events up to 12 months post-procedure | 12 months
  Any anticipated complications of PAE should be recorded on the ROPE Register up to 12 months post-procedure. These include: Local dissection, non-target embolisation, groin haematoma, sepsis, transfusion, TUR syndrome, bladder wall injury, antibiotics needed post-PAE (implying infection), and catheterisation. Patient-reported complications include pain, haematuria, haematospermia, retrograde ejaculation, catheterisation, and hospital re-admission.
IPSS comparison of other treatments (HoLEP, Open prostatectomy) to PAE, 12 months post-procedure | 12 months
  Descriptive statistics for comparison of PAE with other treatments (HoLEP, Open prostatectomy) using IPSS.
IIEF comparison of TURP, HoLEP and Open prostatectomy to PAE, 12 months post-procedure. | 12 months
  Descriptive statistics for comparison of PAE with other treatments (Open Prostatectomy or laser surgery) using IIEF.
Prostate volume comparison of TURP, HoLEP and Open prostatectomy to PAE, 12 months post-procedure. | 12 months
  Descriptive statistics for comparison of PAE with other treatments (TURP, Open Prostatectomy or HoLEP) using prostate volume.
Urinary flow study comparison of TURP, HoLEP and Open prostatectomy to PAE, 12 months post-procedure. | 12 months
  Descriptive statistics for comparison of PAE with other treatments (TURP, Open Prostatectomy or HoLEP) using urinary flow studies.

CONTACTS AND LOCATIONS:
Locations (17):
- United Kingdom (17):
  - Colchester Hospital University NHS Foundation Trust, Colchester, Essex
  - East Kent Hospitals University NHS Foundation Trust, Canterbury, Kent
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - The Royal Bournemouth and Christchurch NHS Foundation Trust, Bournemouth
  - University Hospitals Coventry & Warwickshire NHS, Coventry
  - Frimley Park Hospital NHS Found Trust, Frimley
  - NHS Greater Glasgow and Clyde, Glasgow
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Oxford University Hospitals NHS Trust, Oxford
  - Plymouth Hospitals NHS Trust, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - University Hospital North Staffordshire NHS Trust, Stoke-on-Trent
  - Royal Cornwall Hospitals NHS Trust, Truro

REFERENCES:
- [Result] Ray AF, Powell J, Speakman MJ, Longford NT, DasGupta R, Bryant T, Modi S, Dyer J, Harris M, Carolan-Rees G, Hacking N. Efficacy and safety of prostate artery embolization for benign prostatic hyperplasia: an observational study and propensity-matched comparison with transurethral resection of the prostate (the UK-ROPE study). BJU Int. 2018 Aug;122(2):270-282. doi: 10.1111/bju.14249. Epub 2018 May 6. PMID 29645352
- [Derived] Patel N, Yung N, Vigneswaran G, de Preux L, Maclean D, Harris M, Somani B, Bryant T, Hacking N, Modi S. 1-year cost-utility analysis of prostate artery embolization (PAE) versus transurethral resection of the prostate (TURP) in benign prostatic hyperplasia (BPH). BMJ Surg Interv Health Technol. 2021 Nov 10;3(1):e000071. doi: 10.1136/bmjsit-2020-000071. eCollection 2021. PMID 35047801